CLINICAL TRIAL: NCT00330252
Title: Weekly Subcutaneous Alemtuzumab and Rituximab for Relapsed CLL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Jennifer R. Brown, MD, PhD, Assistant Professor of Medicine, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-404
Record Dates: First submitted 2006-05-25; First posted 2006-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Relapsed Chronic Lymphocytic Leukemia; Alemtuzumab; Campath; Rituximab; Rituxan
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alemtuzumab & Rituximab (Experimental): Alemtuzumab Dosage will vary during Phase I of trial: Given intravenously on days 1, 3, and 5 for weeks one and two, on days 1 and 4 for weeks three and four and on day 1 for weeks five through eight. Participants may receive either one eight-week course of treatment or two eight-week courses of treatment (16 weeks)
  Rituximab- Given intravenously on day 1 of every week for eight weeks (or 16 weeks)
  Interventions: Drug: Rituximab; Drug: Alemtuzumab

INTERVENTIONS:
Drug: Rituximab — Given intravenously on day 1 of every week for eight weeks (or 16 weeks)
Drug: Alemtuzumab — Drug: Alemtuzumab Dosage will vary during Phase I of trial: Given intravenously on days 1, 3, and 5 for weeks one and two, on days 1 and 4 for weeks three and four and on day 1 for weeks five through eight. Participants may receive either one eight-week course of treatment or two eight-week courses of treatment (16 weeks).

SUMMARY:
The purpose of this study is to determine whether the combination of alemtuzumab and rituximab is safe and effective in treating patients with relapsed Chronic Lymphocytic Leukemia (CLL) and to determine whether alemtuzumab can be given as a single weekly subcutaneous dose, together with rituximab.

DETAILED DESCRIPTION:
This study proposes to combine alemtuzumab, which effectively treats peripheral blood and bone marrow disease in CLL, with rituximab, which has activity in lymph node disease, in a streamlined and convenient administration schedule. Preclinical data support synergistic interaction of the two. The primary objectives are (1) to determine the overall and complete response (CR) rate in patients with relapsed CLL and to determine the safety of the combination, and (2) the safety of higher doses of alemtuzumab at less frequent intervals. Secondary objectives are (1) to describe the duration of response, progression-free survival, and overall survival in patients not proceeding to allo transplant, (2) to determine the improvement in overall and complete response associated with administration of a 2nd eight week course of therapy, and (3) to assess minimal residual disease in certain patients and to correlate those results with survival. If at least 16 responses are observed among 35 patients, then the treatment will be considered promising.

The development of antibody therapies has held promise for CLL, since CLL therapies have been palliative, with no established therapy shown to improve survival. Studies have suggested that in contrast to what is seen with fludarabine and alkylating agents, response rates to alemtuzumab are maintained in CLL subjects with P53 mutations. Tolerability of rituximab and its major activity in nodes make it an attractive candidate for combination with alemtuzumab.

This is a single center (DF/HCC), single arm, multi cohort, phase I study, with treatment on an outpatient basis. If the initial alemtuzumab dose of 30 mg sc d1, 3,and 5 is tolerated, there will be dose escalations in cohorts of 3, up to 90 mg d1 per week. Following determination of a maximum tolerated dose, accrual of all remaining patients will occur at that dose. Subjects will be restaged after 8 weeks of therapy, and may proceed to transplant. If deriving benefit, but not in CR, subjects may receive another 8 weeks of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be diagnosed with B-CLL / SLL (B-chronic lymphocytic leukemia / small lymphocytic lymphoma) based on the standard histologic and immunophenotypic criteria described in the WHO classification of lymphoid malignancies, including immunophenotypic confirmation that the tumor cells co-express B cell antigens CD19 / 20 and CD5. Mantle cell lymphoma should be excluded based on positive staining of the tumor cells for CD23, or the absence of staining of the tumor cells for cyclin D1 or the absence of t(11;14).
* The above diagnosis must be confirmed at Brigham & Women's Hospital or Dana-Farber Cancer Institute.
* Subjects must have relapsed after at least one prior fludarabine-containing regimen and require treatment based on NCI-WG criteria (Appendix A).
* Subjects must have measurable disease (lymphocytosis > 5,000 / ml, or palpable lymphadenopathy or CT measurable lymphadenopathy > 1.5 cm, or bone marrow involvement >30%).
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment.
* Age >= 18
* WHO Performance status <= 2
* Subject has provided written informed consent.
* Expected survival > 3 months

Exclusion Criteria:

* History of HIV
* Active infection uncontrolled by appropriate antibacterial, antiviral or antifungal therapy
* Known CNS involvement with CLL
* Pregnant (a negative serum pregnancy test should be performed for all women of childbearing potential within 7 days of treatment) or currently lactating women
* Prior anti-neoplastic therapy within the last three weeks
* Patients will NOT be excluded because they have received prior rituximab or alemtuzumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-05; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of alemtuzumab given once weekly | 2 years
Response rate of combined rituximab and subcutaneous alemtuzumab (complete or partial response) | 2 years

SECONDARY OUTCOMES:
Dose limiting toxicities defined as non-hematologic toxicity of grade 3 or greater or irreversible grade 2 renal, neurologic or cardiac toxicity or infectious toxicities if grade 4 or greater | 2 years
Dose limiting toxicities defined as hematologic toxicities of grade 3 or greater neutropenia or thrombocytopenia for greater than 2 weeks OR ANC < 250 or platelets < 20,000 | 2 years
Response rate as measured by Chest/abdominal/pelvic (+/- neck) CT 4 to 8 weeks following conclusion of 8 Weeks of therapy or at time of study withdrawal | 2 years
Response rate as measured by physical exam of lymph nodes at 4 to 8 weeks following conclusion of 8 Weeks of therapy or at time of study withdrawal, then every 3 months until disease progression | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R Brown, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Brown JR, Messmer B, Werner L, Davids MS, Mikler E, Supko JG, Fisher DC, LaCasce AS, Armand P, Jacobsen E, Dalton V, Tesar B, Fernandes SM, McDonough S, Ritz J, Rassenti L, Kipps TJ, Neuberg D, Freedman AS. A phase I study of escalated dose subcutaneous alemtuzumab given weekly with rituximab in relapsed chronic lymphocytic leukemia/small lymphocytic lymphoma. Haematologica. 2013 Jun;98(6):964-70. doi: 10.3324/haematol.2013.086207. Epub 2013 May 3. PMID 23645694